CLINICAL TRIAL: NCT05575063
Title: Clinical Investigation of Healon EndoCoat Ophthalmic Viscosurgical Device (OVD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VSCO-110-LOKE
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Investigational Healon EndoCoat (Experimental): Eligible subjects to be randomly assigned to receive investigational Healon EndoCoat in one eye and control Healon EndoCoat in fellow eye.
  Interventions: Device: Investigational Healon Endocoat; Device: Control Healon EndoCoat
- Control Healon EndoCoat (Active Comparator): Eligible subjects to be randomly assigned to receive investigational Healon EndoCoat in one eye and control Healon EndoCoat in fellow eye.
  Interventions: Device: Investigational Healon Endocoat; Device: Control Healon EndoCoat

INTERVENTIONS:
Device: Investigational Healon Endocoat — Ophthalmic Viscoelastic device
Device: Control Healon EndoCoat — Ophthalmic Viscoelastic device

SUMMARY:
Prospective, multicenter, paired-eye, randomized, subject/evaluator-masked clinical investigation of the experimental EndoCoat OVD versus the control EndoCoat OVD.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum 22 years of age
2. Cataracts for which extraction and posterior chamber IOL implantation have been planned in both eyes
3. Potential for postoperative best corrected distance visual acuity (BCDVA) of 20/40 Snellen or better
4. Clear intraocular media, other than cataract
5. Availability, willingness and sufficient cognitive awareness to comply with examination procedures
6. Signed informed consent and HIPAA authorization

Exclusion Criteria:

1. Pupil abnormalities (non-reactive, fixed pupils, or abnormally shaped pupils)
2. Recent ocular trauma or ocular surgery that is not resolved/stable or may affect clinical outcomes or increase risk to the subject
3. Prior corneal refractive (LASIK, LASEK, RK, PRK, etc.) or intraocular surgery
4. Subjects with diagnosed degenerative visual disorders (e.g., macular degeneration or other retinal disorders) that are predicted to cause visual acuity losses to a level worse than 20/40 Snellen during the study.
5. Prior, current, or anticipated use during the course of the 3-month study of tamsulosin or silodosin (e.g., Flomax, Flomaxtra, Rapaflo) that may, in the opinion of the investigator, confound the outcome or increase the risk to the subject (e.g., poor dilation or a lack of adequate iris structure to perform standard cataract surgery)
6. Conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration or tilt, such as pseudoexfoliation, trauma, or posterior capsule defects
7. Use of systemic or ocular medications that may affect vision or IOP
8. Corneal abnormalities such as stromal, epithelial or endothelial dystrophies that are predicted to cause visual acuity losses to a level worse than 20/40 Snellen during the study, or in the opinion of the investigator, may confound the outcome(s) of the study
9. Poorly-controlled diabetes
10. Acute, chronic, or uncontrolled systemic or ocular disease or illness that, in the opinion of the investigator, would increase the operative risk or confound the outcome(s) of the study (e.g., immunocompromised, connective tissue disease, suspected glaucoma, glaucomatous changes in the fundus or visual field, ocular inflammation, etc.).
11. Known steroid responder
12. Ocular hypertension of ≥ 20 mmHg, medically-controlled ocular hypertension (regardless of IOP value), or glaucomatous changes in the optic nerve
13. Endothelial cell count (ECC) lower than 1800 cells/mm2 preoperatively (based on the average of the three cell counts as taken by the Konan Specular Microscope)
14. Known ocular disease or pathology that may affect visual acuity or that may be expected to require retinal laser treatment or other surgical intervention during the course of the study (macular degeneration, cystoid macular edema, diabetic retinopathy, etc.)
15. Patient is pregnant, plans to become pregnant, is lactating or has another condition associated with the fluctuation of hormones that could lead to refractive changes
16. Concurrent participation or participation within 60 days prior to preoperative visit in any other clinical trial

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision, Inc. Clinical Trial, Study Director — Johnson & Johnson Surgical Vision, Inc.
Locations (8):
- United States (8):
  - Empire Eye & Laser Center, Bakersfield, California
  - Southern California Eye Physicians and Associates, Long Beach, California
  - Scott & Christie and Associates, Cranberry Township, Pennsylvania
  - Eye Care Specialists, Kingston, Pennsylvania
  - Berkeley Eye Institute, P.A., Houston, Texas
  - Focal Point Vision, San Antonio, Texas
  - Parkhurst NuVision, San Antonio, Texas
  - Virginia Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 165 subjects were enrolled in the study. Of these, 131 subjects (261 eyes) received the treatment and were included in the analysis.
Pre-assignment Details: Participant Flow table and outcome measures arms are divided by 'investigational OVD, one eye treated with investigational HEALON EndoCoat OVD' vs. 'control OVD, one eye treated with control HEALON EndoCoat OVD'.
Units Other Than Participants: Eyes
Groups:
- OVD Groups: Control OVD: One eye treated with control HEALON EndoCoat OVD Investigational OVD: One eye treated with investigational HEALON EndoCoat OVD
Period: Overall Study
Arm/Group | OVD Groups
Started | 131; 261 Eyes
Investigational OVD | 131; 131 Eyes
Control OVD | 130; 130 Eyes
Completed Investigational OVD | 131; 131 Eyes
Completed Control OVD | 129; 129 Eyes
Completed | 130; 260 Eyes
Not Completed | 1; 1 Eyes
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Of the 131 treated subjects, data from 100% (131 /131) of the eyes treated with the investigational OVD and 99.2% (129/130) of the eyes treated with the control OVD were available at the final 3-month visit.
Groups:
- Safety Population: Total of 131: 129 contralaterally treated with investigational and control OVDs; 1 bilaterally treated with the investigational OVD; 1 unilaterally treated with the control OVD
Arm/Group | Safety Population
Number analyzed (Participants) | 131
Age, Customized [Count of Participants; unit: Participants]
  Age Group: <60 years old | 9
  Age Group: 60-69 years old | 58
  Age Group: 70-79 years old | 58
  Age Group: >=80 years old | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 78
  Sex: Male | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 23
  Ethnicity: Not Hispanic or Latino | 108
  Ethnicity: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0
  Race: Asian | 5
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: Black or African American | 9
  Race: White | 111
  Race: More than one race | 6
  Race: Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cumulative IOP Spike Rate From Safety Endpoint
Description: The cumulative IOP spike rate is the proportion of eyes that experienced at least one IOP spike within each arm during the 3-month postoperative period. The status of the cumulative IOP spike is either 'Yes, Spike' or 'No, Non-Spike,' and the results of the cumulative IOP spike rate are presented in percentage. For this outcome measure, subjects have been analyzed as per treated received, which gives investigational OVD of 131 participants and 131 eyes treated; and control OVD of 130 participants and 130 eyes treated.
Time Frame: 3-month postoperative
Population: Percentage cumulative IOP spike rate
Measure: Number; unit: Percentage
Units Other Than Participants: Eyes
Groups:
- Investigational OVD: One eye with investigational HEALON EndoCoat OVD
- Control OVD: One Eye with control HEALON EndoCoat OVD
Arm/Group | Investigational OVD | Control OVD
Number analyzed (Participants) | 131 | 130
Number analyzed (Eyes) | 131 | 130
Percentage | 7.54 | 7.46
Statistical Analysis 1: Comparison: Investigational OVD vs Control OVD; Test type: Non-Inferiority — All analyzed numbers are in percentage. The success criterion for the primary safety endpoint was met (Safety Population), as the investigational device (HEALON EndoCoat OVD) demonstrated non-inferiority to the control device (HEALON EndoCoat OVD) with respect to the difference in IOP spike rate, estimated to be 0.08% (with the 95% confidence interval of [-5.07%; 5.23%]); Mixed Models Analysis; Not Measured = 0.08, 95% CI 2-sided [-5.07 to 5.23], Standard Error of Mean 2.63 — All values in this section are in percentage

2. Primary Outcome: ECC Percent Change From Effectiveness Endpoint
Description: The success criterion for the primary effectiveness endpoint was met (modified ITT Population) as the investigational device (HEALON EndoCoat OVD) demonstrated non-inferiority to the control device (HEALON EndoCoat OVD) with respect to the difference in mean ECC percent change. For this outcome measure, subjects have been analyzed as per planned randomization schema, which gives investigational OVD of 130 participants and 130 eyes randomized; and control OVD of 131 participants and 131 eyes randomized.
Time Frame: 3-month postoperative
Population: ECC Change in Percentage in Negative number value
Measure: Mean (Standard Error); unit: Percentage Change
Units Other Than Participants: Eyes
Arm/Group | Investigational OVD | Control OVD
Number analyzed (Participants) | 130 | 131
Number analyzed (Eyes) | 130 | 131
Percentage Change | -9.03 (1.31) | -8.53 (1.27)
Statistical Analysis 1: Comparison: Investigational OVD vs Control OVD; Test type: Non-Inferiority — All analyzed numbers are in percentage. The success criterion for the primary effectiveness endpoint was met (modified ITT Population) as the investigational device (HEALON EndoCoat OVD) demonstrated non-inferiority to the control device (HEALON EndoCoat OVD) with respect to the difference in mean ECC percent change, estimated to be -0.50% (with the 95% confidence interval of [-3.37%; 2.37%]); Mixed Models Analysis; Difference in Percent Change = -0.5, 95% CI 2-sided [-3.37 to 2.37], Standard Error of Mean 1.46 — All values are in percentage

ADVERSE EVENTS:
Time Frame: 3 months postoperative follow-up
Description: There were a total of 32 AEs.
Groups:
- Investigational OVD: One eye treated with investigational HEALON EndoCoat OVD
- Control OVD: One Eye Treated with control HEALON EndoCoat OVD
Arm/Group | Investigational OVD | Control OVD
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/130
Serious Adverse Events (participants affected / at risk) | 14/131 | 17/130
Other Adverse Events (participants affected / at risk) | 0/131 | 0/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational OVD (N=131) | Control OVD (N=130)
Increased IOP (Eye disorders) | 11 (11) | 11 (11)
Cystoid Macula Edema (Eye disorders) | 2 (2) | 2 (2)
Central Serous Retinopathy (Eye disorders) | 1 (1) | 1 (1)
Retained Lens Material (Eye disorders) | 0 (0) | 1 (1)
Residual Refractive Error (Eye disorders) | 0 (0) | 1 (1)
Hospitalization due to chest pain (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT05575063/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT05575063/SAP_001.pdf